CLINICAL TRIAL: NCT03279276
Title: Selection of Hip Prosthesis for Younger Patients? Primoris® Short Femur Component vs. Echo® Standard Femur Component. Comparison of Bone Re-modeling, Prosthetic Migration and Gait Function. Controlled Randomized Study of 60 Patients.
Brief Title: Selecting the Right Hip Prosthesis for Young Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20170030
Record Dates: First submitted 2017-08-31; First posted 2017-09-12 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Hip
Keywords: Hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primoris (Experimental): Total hip arthroplasty surgery using a Primoris® femur component, Exceed ® acetabular cup + E-poly liner ®.
  Interventions: Procedure: Total Hip Arthroplasty
- Echo (Active Comparator): Total hip arthroplasty surgery using a standard uncemented Echo® femur component, Exceed ® acetabular cup + E-poly liner ®.
  Interventions: Procedure: Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Total Hip Arthroplasty — The usual procedures of the department: Moore incision and insertion of uncemented joints (exceed with vitamin E enriched polyethylene liner and 32 or 36 mm head). Cyclokaprone is administered peroperatively (bleeding-reducing), antibiotics and thrombosis prophylaxis. Follow the usual rehabilitation regimes, fast track, incl. Use of crutches and must support within the pain limit, possibly with crutches the first 4 weeks after surgery, then full load.
  By default, postoperative X-ray and RSA recordings will be performed on the 1st or 2nd postoperative day. The surgery will be performed by specialist physicians in orthopedic surgery associated with the hip arthroplasty sector.

SUMMARY:
There have been no previously published clinical randomized studies comparing Primoris®, short stem, hip prosthesis with standard uncemented hip arthroplasty in relation to bone density and function development. This is the subject for this study.

DETAILED DESCRIPTION:
The overall purpose of this study is to show whether the Primoris® hip prosthesis results in a smaller loss of bone density than standard hip prosthesis, which in the longer term may result in an improved survival of prosthesis No. 2 after revision / replacement of a Primoris® hip prosthesis.

The primary outcome is periprosthetic bone quality in Primoris® hip prosthesis compared to standard hip prosthesis measured by DXA scanning.

The secondary outcomes are to assess:

1. The hip function measured by gait analysis.
2. Hip strength at pressure gauge.
3. Prosthetic migration / migration measured by radio-stereometric analysis (RSA).
4. Patient satisfaction measured by PROMs.

ELIGIBILITY:
Inclusion Criteria:

Women ≤ 45 years or men ≤ 55 years with hip osteoarthritis, suitable for hip prosthesis.

Patients who wish to participate in the project and give written consent after oral and written information.

Exclusion Criteria:

1. Patients with previous bone disease, metabolic disease, including diabetes, or the use of drugs that affect bone density.
2. Smoking more than 20 cigarettes daily
3. Patients with fracture in the femur or acetabulum.
4. Patients who do not understand the given patient information
5. Competing disorder requiring treatment with antiinflammatory drugs (NSAIDs, steroid, cytostatics).
6. Estimated residual life <10 years
7. Rheumatoid arthritis or other arthritis (eg psoriasis arthritis).
8. Previous surgery on the relevant hip joint.
9. Co-Morbidity (ASA Group 3-5).
10. Neurological disorder that compromises motor skills and rehabilitation.
11. Pregnancy.
12. Osteoarthritis secondary to mb. Calvé-Legg-Perthes / Avascular Caput Necrosis, Epiphysiolysis Capitis Femoris and Multiple Epiphysic Dysplasia.
13. Acetabular dysplasia with secondary subluxation (Crowe grade II to IV).
14. Previously detected osteoporosis or osteoporosis detected by current DXA scanning.
15. Ongoing treatment with osteoporosis medicine (bisphosphonates, estrogen receptor modulators and parathyroid hormone, etc.).
16. Aseptic caput necrosis (posttraumatic, idiopathic).
17. Varus or valgus deformity in proximal femur (collum angle <125 ° or> 145 °.)
18. Collum femoris assessed too retro- or anteverted.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density | 2 -10 years
  Bone density around the prosthesis measured by serial Dual X-ray Absorptiometry (DXA) scans.

SECONDARY OUTCOMES:
Gait analysis | 1 year
  Walking function measured by gait analysis and hip strength at dynamometer test pre and 12 months postoperatively.
Radio Stereometric Analysis (RSA) | 2-10 years
  Prosthetic migration / migration measured by X-ray Radio-stereophotogrametic-analyzes
European Quality of life in 5 Dimensions (EQ5D) | 2-10 years
  This is a well defined Patient Reported Outcome Measure (PROM) that doesn't need further explanation.
Harris Hip Score (HHS) | 2-10 years
  This is a well defined Patient Reported Outcome Measure (PROM) that doesn't need further explanation.
Oxford Hip Score (OHS), | 2-10 years
  This is a well defined Patient Reported Outcome Measure (PROM) that doesn't need further explanation.
University of California Los Angeles Activity Score (UCLA) | 2-10 years
  This is a well defined Patient Reported Outcome Measure (PROM) that doesn't need further explanation.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 2-10 years
  This is a well defined Patient Reported Outcome Measure (PROM) that doesn't need further explanation.
Forgotten Joint Score (FJS) | 2-10 years
  This is a well defined Patient Reported Outcome Measure (PROM) that doesn't need further explanation.

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Laursen, MD, PhD, Principal Investigator — Northern ODD
Locations (1):
- Northern Orthopaedic Division, Clinic Farsø, Aalborg University Hospital, Farsø, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No